CLINICAL TRIAL: NCT04819048
Title: Efficacy of Acupuncture and Low-Level Laser in Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP2021-12-10202
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Low-Level Laser Therapy; acupuncture
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Laser Therapy+acupuncture (Experimental): The laser light will be applied in 6 points on the affected side: anterior to the mandibular condyle and intraauricular toward the temporomandibular joint; 2 points irradiation on the superficial masseter muscle and 2 points on the anterior temporal muscle bundle. Each point will be irradiated for 30 seconds for a total of 180 seconds.
  After LLLT irradiation,the following acupuncture points will be selected: Jiache,Xiaguan,Quanliao,Baihui,Fengchi, Hegu.The needles will be inserted and rotated manually with a frequency of about 100 turns per minute clockwise and counterclockwise ,as above vertically into a depth of 25-30 mm to achieve the proper feel called "Deqi" in every point on the affected side, and then the needles will be retained for 30 minutes.
  Interventions: Device: Low-Level Laser Therapy+acupuncture
- Low-Level Laser Therapy (Active Comparator): The laser light will be applied in 6 points on the affected side: anterior to the mandibular condyle and intraauricular toward the temporomandibular joint; 2 points irradiation on the superficial masseter muscle and 2 points on the anterior temporal muscle bundle. Each point will be irradiated for 30 seconds for a total of 180 seconds.
  Interventions: Device: Low-Level Laser Therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy+acupuncture — The experimental group will be firstly irradiated by the GaAlAs infrared laser (CDHC,Denlase 980/7 Diode Laser Therapy System,China), with an output of 500 mW, emitting radiation wavelength of 980 nm, spot size 0.2cm2 ,15J/point, in a continuous mode .The therapeutic LLLT application is achieved through direct contact of the probe on the skin.
  The needles using are disposable, sterile, individually packed, and made of stainless steel (Hua Tuo; Suzhou Medical Supplies Factory Co, Ltd,Suzhou, China), in sizes 0.25 mm ×40 mm.Asepsis of the skin will be performed with cotton wool and 75% alcohol.
  Arms: Low-Level Laser Therapy+acupuncture
Device: Low-Level Laser Therapy — The experimental group will be firstly irradiated by the GaAlAs infrared laser (CDHC,Denlase 980/7 Diode Laser Therapy System,China), with an output of 500 mW, emitting radiation wavelength of 980 nm, spot size 0.2cm2 ,15J/point, in a continuous mode .The therapeutic LLLT application is achieved through direct contact of the probe on the skin.
  Arms: Low-Level Laser Therapy

SUMMARY:
Temporomandibular joint disorders (TMD) , a musculoskeletal condition , includes a series of clinical problems involving the temporomandibular joint (TMJ), the masticatory muscles, and related structures.This study evaluates the efficacy of integrated traditional Chinese and western medicine in the treatment of TMD.

DETAILED DESCRIPTION:
In this study, 84 patients ranging in age from 18 to 65 years with diagnoses of TMD will be randomly divided into two groups: an experimental group (EG) who will receive the integrated traditional Chinese and western medicine treatment group(with Low-Level Laser Therapy+acupuncture) and a control group who will receive the only western medicine treatment(with Low-Level Laser Therapy).Both approaches will be applied 3times a week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of TMD according to the Diagnostic Criteria for TMD Research Diagnostic Criteria (DC/TMD）which are manifested as joint pain during mouth opening and chewing, mouth opening limitation (<40mm), joint clanging, masticatory creatine distension and weakness, which affects normal eating.
2. Aged 18-65;
3. Unilaterally;
4. No any other treatment on TMD in the last 3 months;

Exclusion Criteria:

1. there are tumors, joint degeneration and other serious lesions ;
2. Patients with a history of TMJ trauma or surgery,joint anatomical variation;
3. women pregnant and suckling period;
4. serious systemic diseases of bone and joint, such as rheumatoid arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | Change from baseline Visual analogue scale at week 3
  TMD pain will be quantified by the VAS, which is a 10-cm line ranging from 0 cm (no pain at all) to 10 cm (the worst possible pain). The patients are instructed to choose the grade of their spontaneous pain intensity on the 10 points scale during resting, mouth opening, and chewing.And then the operator takes the maximum from that.

SECONDARY OUTCOMES:
Tempommandibular Opening Index(TOI) | Change from baseline Tempommandibular Opening Index at week 3
  TOI=(Maximum voluntary opening-passive opening)/Maximum voluntary opening+Passive opening)× 100％.
  The maximum mouth opening without pain will be recorded by placing a millimeter ruler in a vertical position, from the incisal edge of the maxillary left central incisor to the incisal edge of the mandibular left central incisor.
  Based on the the maximum opening, the researcher uses thumb and forefinger slowly against the upper and lower incisor , with soft and stable pressure until the distance no longer increases .This is called the passive opening .

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Integrated Traditional Chinese and Western Medicine, Beijing, Beijing Municipality, China